CLINICAL TRIAL: NCT00369252
Title: A Phase I Study of TheraCIM-hR3 (YMB1000) in Patients With Solid Tumours
Brief Title: Phase I Study of Nimotuzumab in Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Collaborators: CIMYM BioSciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMB1000-007
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Advanced and/or Metastatic Solid Tumours
Keywords: Nimotuzumab; TheraCIM; H-R3; Solid tumours; EGFR; Monoclonal antibody
MeSH Terms: interventions — nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab (TheraCIM h-R3)

SUMMARY:
This is a phase I trial of nimotuzumab that will be conducted in patients with advanced incurable solid tumors. This is a dose-seeking study to determine the maximum tolerated and recommended phase II doses of nimotuzumab that can be safely given to patients with advanced and/or metastatic solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose-escalating, phase I trial of nimotuzumab in patients with advanced incurable solid tumors. The objective of this study is to determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of nimotuzumab that can be given in a weekly schedule in patients with advanced and/or metastatic solid tumor cancer. This study will also examine the safety, pharmacodynamics and preliminary efficacy of nimotuzumab in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Advanced and/or metastatic solid tumors, refractory to standard curative therapy, or for which no curative therapy exists.
* Clinically or radiologically documented disease. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan.
* Archival tumor specimens evaluable for expression of the EGFR (but EGFR positivity is not a requirement for study entry).
* Patients must have tumor lesions accessible for biopsy for correlative studies. In cases where there are medical contraindications to tumor biopsies, exceptions may be made upon discussion with the Principal Investigators.
* Age > 18 years.
* ECOG performance status of 0,1,2.
* Previous therapy: Previous chemotherapy, hormonal therapy, radiation and/or surgery is permitted with certain restrictions as outlined in the protocol.
* Hematology and chemistry lab results within specifications outlined in the protocol.
* Willingness to give written informed consent.
* Patients must be accessible for treatment and follow-up.
* Protocol treatment is to begin within 2 working days of patient registration.

Exclusion Criteria:

* Pregnant or lactating women. Both men and women enrolled on study should be using adequate birth control measures throughout the course of the study.
* History of second malignancy who have a disease-free interval of less than two years (except cervical cancer in situ or nonmelanomatous skin cancer).
* Untreated brain or meningeal metastases. Patients with treated and stable brain metastases are eligible providing that they have radiologic evidence of disease stabilisation of at least 3 months duration and are asymptomatic.
* Untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction.
* Active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Prior therapy with EGFR targeting therapies, including monoclonal antibodies or small molecule tyrosine kinase inhibitors.
* Allergy to the antibody.
* Concurrent treatment with other experimental drugs or anti-cancer therapy.
* Inability or unwillingness to give written, informed consent prior to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, MD, Principal Investigator — University Health Network, Toronto; Lillian Siu, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada